CLINICAL TRIAL: NCT02076048
Title: LCPUFA Supplementation: A Multi-Modality Imaging Study
Status: Completed | Type: Observational
Sponsor: Kathleen Gustafson, Ph.D. (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor-Investigator, Kathleen Gustafson, Ph.D., Research Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: LCPUFA Supplementation
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Child Development
Keywords: LCPUFA supplementation; Brain Imaging; MRI; MEG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cheek swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Previous LCPUFA Supplementation: Children between the ages of 7 and 10 that were previously enrolled in a study of supplemented LCPUFA formula.

SUMMARY:
The purpose of this study is to take images of the brain in order to see if long-chain polyunsaturated fatty acid (LCPUFA) exposure during infancy influences brain structure and function in middle childhood.

DETAILED DESCRIPTION:
LCPUFAs are essential fatty acids that are found in all cells of the body, particularly in the brain, retina and other nervous tissue. LCPUFAs are found naturally in seeds, nuts, fish and human breast milk. The body can also make LCPUFAs from shorter-chain fatty acid precursors.

The researchers in the study have previously found that LCPUFA supplementation during infancy has a beneficial effect on vision and development in the early years of life. However, researchers feel there is a growing need to better understand if there are structural and/or functional changes in the brain that explain these benefits. It is also important to understand if changes in development are still present later in childhood.

ELIGIBILITY:
Inclusion Criteria:

* Parents consent for children and children have the ability to assent
* Participation as an infant in the original study

Exclusion Criteria:

* Those with orthodontic braces or extensive dental work that would make them unable to have an MRI

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects who were originally enrolled as infants will be invited to participate in the longitudinal follow up study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Event-Related Field (ERF) Amplitude and Latency | Within 1 year post enrollment
  We will use an MEG Event-Related Field (ERF) to study the development of children's cognitive capabilities. The waveform components associated with information processing and response inhibition will be measured in order to assess the developmental progress of LCPUFA effects with increasing age.
Regional gray and white matter brain volume | Within 1 year post enrollment
  Structural brain imaging is widely used to measure gray and white matter maturation patterns in young children. We will use automated, sensitive, and validated methods to test whether LCPUFA supplementation positively impacts changes in the brain associated with higher functioning and intelligence.

SECONDARY OUTCOMES:
Identify structural and metabolic mediators | Within 1 year post enrollment
  In a single imaging session, we will measure metabolic biomarkers associated with cellular mechanisms such as bioenergetics, membrane status, and oxidative state, each of which have been implicated as associated with LCPUFA supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Gustafson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Lepping RJ, Honea RA, Martin LE, Liao K, Choi IY, Lee P, Papa VB, Brooks WM, Shaddy DJ, Carlson SE, Colombo J, Gustafson KM. Long-chain polyunsaturated fatty acid supplementation in the first year of life affects brain function, structure, and metabolism at age nine years. Dev Psychobiol. 2019 Jan;61(1):5-16. doi: 10.1002/dev.21780. Epub 2018 Oct 11. PMID 30311214